CLINICAL TRIAL: NCT07063082
Title: Efficacy Of Erythromycin Phonophoresis on Chronic Rhinosinusitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, nahla mahmoud mohamed elkassas, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/005150
Record Dates: First submitted 2025-05-30; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Chronic Rhinosinusitis
Keywords: Erythromycin; Phonophoresis; ultrasound
MeSH Terms: interventions — Ultrasonography; Erythromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Erythromycin Phonophoresis + Medical treatment (Experimental): This group will include 30 patients with chronic rhinosinusitis who will receive Erythromycin phonophoresis 12 session, 3 days per week, and medical treatment (saline nasal wash) 3 times daily for a month.
  Interventions: Other: Erythromycin Phonophoresis; Other: Medical treatment
- Ultrasound + Topical Erythromycin + Medical treatment (Active Comparator): This group will include 30 patients with chronic rhinosinusitis who will receive ultrasound followed by topical use of Erythromycin gel on nose 12 session , 3 days per week and medical treatment (saline nasal wash) 3 times daily for a month.
  Interventions: Device: Ultrasound (US); Drug: Topical Erythromycin; Other: Medical treatment
- Medical treatment (Other): This group includes 30 patients with chronic rhinosinusitis who will receive their medical treatment (saline nasal wash) 3 times daily for a month
  Interventions: Other: Medical treatment

INTERVENTIONS:
Other: Erythromycin Phonophoresis — The procedures of ultrasound phonophoresis will be as follows: Patients will be positioned comfortably, sitting in a relaxed position. The physiotherapist will explain the treatment procedures to the patient. The device cables will be checked before each session. The treatment will last 5 minutes for each maxillary sinus. The frequency will be set to 1 MHz, and the intensity will be 1 W/Cm2 for the maxillary sinuses. The ultrasound will be pulsed, and the treatment will consist of 12 sessions, 3 days per week.
  Arms: Erythromycin Phonophoresis + Medical treatment
Device: Ultrasound (US) — Therapeutic US is produced by a transducer composed of a piezoelectric crystal, which converts electric energy into alternating compression and rarefaction of sound waves at a frequency greater than 20 kHz. The amplitude of the US wave is proportional to the displacement of the US transducer head during each half cycle. The amplitude represents the wave energy.
  The ultrasound waves penetrate the tissue on the way to the target organ and have two mechanisms of action (thermal and non-thermal), which may potentially work synergistically to reduce nasal symptoms (nasal blockage and secretions).
  Arms: Ultrasound + Topical Erythromycin + Medical treatment
Drug: Topical Erythromycin — Erythromycin is a 14-member macrolide originally discovered in the 1950s. It has broad-spectrum antimicrobial action, inhibiting bacterial protein synthesis. studies have shown that erythromycin has immunomodulatory and anti-inflammatory activity independent of its antimicrobial action Erythromycin is a broad-spectrum macrolide antibiotic, wherein its bactericidal effect occurs by the inhibition of protein synthesis. It is used for the treatment of infections affecting the skin and mucosa; it shows immunomodulatory characteristics
  Other Names: Erythromycin
  Arms: Ultrasound + Topical Erythromycin + Medical treatment
Other: Medical treatment — Saline nasal wash 3 times daily for a month.

SUMMARY:
The purpose of the study is to evaluate the therapeutic effect of erythromycin phonophoresis in reducing chronic rhinosinusitis.

DETAILED DESCRIPTION:
Chronic rhinosinusitis (CRS) is defined as "inflammation of the nose and the paranasal sinuses characterized by two or more symptoms, one of which should be either nasal blockage, obstruction, congestion or nasal discharge (anterior or posterior nasal drip) with/without facial pain or pressure, reduction or loss of smell, endoscopic signs of nasal polyps, mucopurulent discharge primarily from middle meatus, oedema, mucosal obstruction primarily in middle meatus and computed tomography (CT) changes (mucosal changes within the osteomata complex and/or sinuses)".

CRS may be a benign disorder, but it has significant morbidity. If not treated, the quality of life is poor. The condition is known to exacerbate asthma and can even lead to meningitis and brain abscess formation- which increases morbidity and mortality. Patients with chronic sinusitis who are treated usually have satisfactory outcomes. Symptom relief can be obtained after functional endoscopic sinus surgery in about 75% of patients who fail to respond to medical management. In rare cases, chronic sinusitis can result in orbital and intracranial infections, leading to visual and neurological deficits.

This study will design to provide a guideline about effect of erythromycin phonophoresis on chronic rhinosinusitis and to assist in planning ideal treatment program.

The treatment for chronic rhinosinusitis is realized through the use of medications such as corticosteroids, antibiotics and antimycotics or surgical procedures. However, treatments are not always effective, which makes patients adhere to other therapeutic modalities, including medicinal herbs, homeopathy and probiotics. A modality that stands out is the use of therapeutic ultrasound, which has shown promising results for its anti-inflammatory and antinociceptive activity.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 25-50 years.
* Male and female patients will participate in the study.
* All patients have chronic rhinosinusitis.
* All patients enrolled in the study will have their informed consent.
* CT will include at least affection of maxillary sinus.

Exclusion Criteria:

* Patients with pacemaker
* Patients diagnosed with cancer.
* Pregnant women
* Patients with impaired vascular circulation
* Patients who suffer from mental or psychological disorders.
* Patients with any systemic diseases that may interfere with the objectives of the study.
* Congenital defects on face and nose.
* Fracture of nose or face.
* Polypoidal patients.
* Allergic patients.
* Previous nasal surgery.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-07-07 (Estimated); Primary Completion 2025-09-07 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Sinusitis symptom score (SSS) | one month
  Sinusitis Symptom Scores will be based on a visual analogue scale (VAS) well established. In this method, the six symptoms will be assessed using a scale of 0±10, where zero represents no symptom and 10 represents the most severe symptom imaginable

SECONDARY OUTCOMES:
Computerized tomography scan (CTS) | one month
  CT scan (TOSHIBA, MODEL TSX-035A, INPUT POWER 50kVA), will assess the mucosal thickening of maxillary sinuses

CONTACTS AND LOCATIONS:
Overall Officials: Nahla Mahmoud Elkassas, B.Sc, Principal Investigator — Physotherapist at Alexanderia Police Hospital; Hussein Gamal Hussein Mogahed, PhD, Study Chair — Assistant Professor, Cairo university; Mustafa Mohamed Abdelnaby, PhD, Study Director — Assistant Professor, Alexandria university; Aya Gamal Fawzy Elsayed, PhD, Study Director — Lecturer, Cairo university
Locations (1):
- Alexanderia Police Hospital, Alexandria, Egypt